CLINICAL TRIAL: NCT00621595
Title: The Effects of Breakfast on Cognitive Functioning
Brief Title: The Effects of Breakfast on Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: R. Terry Pivik, Ph.D. / Principal Investigator, University of Arkansas for Medical Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06278
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: School Breakfast; Diet; Nutrition; Brain Function; Cognition; USDA; Healthy Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Fasting
  Interventions: Dietary Supplement: USDA School Breakfast

INTERVENTIONS:
Dietary Supplement: USDA School Breakfast — Breakfast containing 340 calories, 57 g carbohydrate, 14 g protein, 6 g fat.

SUMMARY:
To test cognitive abilities of 8-11 year old children under conditions of fasting or receiving a full school breakfast.

ELIGIBILITY:
Inclusion Criteria:

* 8-11 years old
* Between 25th and 95th percentile, BMI-for-age

Exclusion Criteria:

* food allergies or some intolerances
* uncorrected vision
* IQ < 80
* Other chronic conditions thought to interfere with the study as determined by the investigator

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2000-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Terry Pivik, Ph.D., Principal Investigator — University of Arkansas for Medial Science
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States